CLINICAL TRIAL: NCT01860560
Title: Effect of High Flow Nasal Cannula (Flowrest®) on Mild-Moderate Sleep Disordered Breathing: A Non-Inferiority Study Versus Nasal Continuous Positive Airway Pressure (CPAP) Therapy
Brief Title: Non-Inferiority Trial of Acute HFT Versus nCPAP
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: this was an error. Study never initiated
Sponsor: Vapotherm, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: RP-HFR2013001Reg
Record Dates: First submitted 2013-05-16; First posted 2013-05-22 (Estimated); Last update posted 2023-05-03 (Actual); Status verified 2023-04

CONDITIONS: Mild-Moderate Obstructive Sleep Disordered Breathing
Keywords: OSA; Obstructive Sleep Apnea; High Flow Therapy; CPAP; HFT; Continuous Positive Airway Pressure; Mild OSA; Moderate OSA
MeSH Terms: conditions — Sleep Apnea, Obstructive | interventions — Continuous Positive Airway Pressure

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- CPAP First / HFT Second (Experimental): Subjects to receive both therapies, order-randomized to receive Continuous Positive Airway Pressure (CPAP) therapy study first, followed by a washout period, and a follow-on High-Flow Therapy (HFT) therapy study
  Interventions: Device: High-Flow Therapy; Device: Continuous Positive Airway Pressure
- HFT First / CPAP Second (Experimental): Subjects to receive both therapies, order-randomized to receive High-Flow Therapy (HFT) therapy study first, followed by a washout period, and a follow-on Continuous Positive Airway Pressure (CPAP) therapy study.
  Interventions: Device: High-Flow Therapy; Device: Continuous Positive Airway Pressure

INTERVENTIONS:
Device: High-Flow Therapy — Blower-based High Flow Therapy delivered by nasal cannula
  Other Names: Vapotherm Flowrest High Flow Therapy
Device: Continuous Positive Airway Pressure — CPAP Therapy delivered by laboratory Positive Airway Pressure titration device.
  Other Names: Respironics Synchrony Lab

SUMMARY:
Order randomized crossover non-inferiority study evaluating the acute efficacy of High Flow Therapy (HFT) as compared to nasal Continuous Positive Airway Pressure therapy (CPAP) in the management of apnea / hypopnea index (AHI).

DETAILED DESCRIPTION:
Study to evaluate the acute efficacy of a single night of High Flow Therapy (HFT) to treat mild-moderate predominantly obstructive Sleep Disordered Breathing, as compared to nasal Continuous Positive Airway Pressure (CPAP) therapy. Subjects will be order-randomized to receive HFT or CPAP in the laboratory, undergo a washout period, and return for the alternative therapy in the laboratory. The hypothesis is that HFT will be non-inferior to CPAP in controlling Apnea/Hypopnea events in this subject set during this study.

Primary outcome will be Apnea / Hypopnea Index (AHI) change on therapy as compared to baseline diagnostic polysomnography.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age
* Previous diagnosis of primarily obstructive mild-moderate Sleep Disordered Breathing during in-laboratory polysomnography
* Ability to read and understand English Language
* Ability to provide informed consent

Exclusion Criteria:

* Unstable medical illness within the last month (30 days)
* Acute / recent upper airway infection
* Prior use of non-continuous positive airway pressure medical technology therapies prescribed by a physician for the management of obstructive sleep disordered breathing (e.g., Provent®, Winx™, mandibular advancement oral appliances, etc.)
* Prior use or exposure to CPAP / Bi-Level / or other non-invasive ventilatory modalities
* Craniofacial or other anatomical anomalies that may predispose patients to upper airway obstruction, or obvious blockage to nasal air flow
* Patients using opioids or amphetamines will be excluded from the study.
* Enhanced oxygen requirement (i.e., FiO2>0.21)
* Patients requiring Bi-Level therapy upon CPAP titration attempt
* Surgery since the diagnostic PSG
* Significant recent sedative/hypnotic use likely, in the opinion of the principle investigator, to impair ventilatory control or impact the subsequent titration of either CPAP therapy or Flowrest therapy (including benzodiazepines, antihistamines, imidazopyridines)
* Significant use of stimulant medications likely, in the opinion of the principle investigator, likely to alter ventilatory or upper airway control and impact the subsequent titration of either CPAP therapy or Flowrest therapy (including amphetamines, high dose caffeine, etc.)
* Significant neurologic or cardiac pathology likely to seriously impact respiratory effort or ventilatory control (e.g., post CVA with ventilatory impairment)
* Presence of significant sleep disorders likely to induce hypersomnolence or interfere with the ability to titrate CPAP therapy or Flowrest therapy (including narcolepsy, PLMS/RLS, severe chronic insomnia, non-OSA obesity hypoventilation syndrome, etc.)
* Unsuitable for inclusion in the opinion of the investigators

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2013-05; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
AHI Change (Therapy v Baseline) | Acute - single night therapy exposure
  Evaluate the change in AHI from baseline for HFT v CPAP therapy

SECONDARY OUTCOMES:
Pulse Oxygen Saturation | Acute single night therapy exposure
  Evaluate the mean, absolute minimum, absolute event-related nadir and mean nadir of pulse oxygen saturation during therapeutic polysomnography of HFT v CPAP
Sleep Architecture (WASO, %W, N1, N2, N3, REM, SL, RL, AI) | Acute single night therapy exposure
  Evaluate changes in sleep architecture on HFT and CPAP therapy as compared to baseline diagnostic polysomnography. Specifically, evaluate any difference between the therapies on %Wake Time (of SPT), % time in stages N1, N2, N3, REM (of TST), Minutes of Wake After Sleep onset, Sleep latency and REM Latency. Any difference in overall non-respiratory arousal index will be assessed.
Respiratory Event Related Arousals | Acute single night therapy exposure
  Compare the incidence of RERA on HFT and CPAP therapy as compared to diagnostic polysomnography.
Respiratory Disturbance Index (RDI) | Acute single night therapy exposure
  Evaluate the RDI on HFT v CPAP therapy as compared to the diagnostic polysomnography.

CONTACTS AND LOCATIONS:
Overall Officials: George Dungan, MPhil Med, Study Director — Vapotherm, Inc.
Locations (1):
- Sleep Disorders Centers of the Mid-Atlantic, Glen Burnie, Maryland, United States